CLINICAL TRIAL: NCT05148364
Title: How Pain Resilience and Spiritual Health Affect the Pain Experience in Patients With Low Back Pain
Brief Title: Pain Resilience and Spiritual Health in Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 211102
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: spirituality; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: interview — A spiritual consultant and a psychologist will interview the participants about their experiences of chronic low back pain, how they interpret their pain experience and how they cope with the persistent pain. Each participant will be interviewed individually.
  Questions related to the following three aspects will be asked:
  1. Attributes: describe the changes in your personality, mood, and general happiness you have observed after you starting having chronic low back pain.
  2. Pain resilience: How would you describe this persisting pain experience? How do you arrange your daily activity? What do you do to deal with this persistent pain?
  3. Spirituality: As a person with chronic low back pain, how do you interpret this pain experience? Do you seek connections with higher powers (such as powers from religion) when you are desperate because of pain? Since the pain is chronic and persistent, it might not go away, how would you define your life?

SUMMARY:
In the management of chronic pain, it is very important to reaffirm the patient's self-worth and ability through psychological support and spiritual care. The role of spiritual consultant is to provide spiritual consultation and spiritual care, so that the medical team can truly implement a whole-person care of the patient including the body, mind, and family. Pain resilience of chronic pain patients' has been found to be a different construct from the general resilience in the field of chronic diseases. Pain resilience emphasizes the cognitive/emotional positivity and behavior persistence of pain patients' when facing pain. So far, there has been no research on the theme of "pain resilience and spiritual health". Researchers have seen the necessity of care and assistance for patients with chronic low back pain. Hence, this study would like to explore "how pain resilience and spiritual health affect the pain experience of patients with chronic low back pain ".

Research objectives: 1. To understand how spiritual health and pain resilience interact to influence the the pain experience in patients with chronic low back pain and 2. To understand how spiritual health and pain resilience interact and influence they way how patients with chronic low back pain cope with pain.

Method: This research plan will be implemented upon obtaining the approval from IRB. An estimated 15 cases will be enrolled. Through in-depth interviews and collection of observational data during interviews, the interviewer will record, transcribe and analyze the narratives and experience descriptions.

The results of this study can become an important basis for clinical care of patients with chronic low back pain.

DETAILED DESCRIPTION:
In the management of chronic pain, it is very important to reaffirm the patient's self-worth and ability through psychological support and spiritual care. The role of spiritual consultant is to provide spiritual consultation and spiritual care, so that the medical team can truly implement a whole-person care of the patient including the body, mind, and family. Pain resilience of chronic pain patients' has been found to be a different construct from the general resilience in the field of chronic diseases. Pain resilience emphasizes the cognitive/emotional positivity and behavior persistence of pain patients' when facing pain. So far, there has been no research on the theme of "pain resilience and spiritual health". Researchers have seen the necessity of care and assistance for patients with chronic low back pain. Hence, this study would like to explore "how pain resilience and spiritual health affect the pain experience of patients with chronic low back pain ".

Research objectives: 1. To understand how spiritual health and pain resilience interact to influence the the pain experience in patients with chronic low back pain and 2. To understand how spiritual health and pain resilience interact and influence they way how patients with chronic low back pain cope with pain.

Method: This research plan will be implemented upon obtaining the approval from IRB. An estimated 15 cases will be enrolled. Through in-depth interviews and collection of observational data during interviews, the interviewer will record, transcribe and analyze the narratives and experience descriptions.

A spiritual consultant and a psychologist will interview the participants about their experiences of chronic low back pain, how they interpret their pain experience and how they cope with the persistent pain. Each participant will be interviewed individually.

Questions related to the following three aspects will be asked:

1. Attributes: describe the changes in your personality, mood, and general happiness you have observed after you starting having chronic low back pain.
2. Pain resilience: How would you describe this persisting pain experience? How do you arrange your daily activity? What do you do to deal with this persistent pain?
3. Spirituality: As a person with chronic low back pain, how do you interpret this pain experience? Do you seek connections with higher powers (such as powers from religion) when you are desperate because of pain? Since the pain is chronic and persistent, it might not go away, how would you define your life?

Plan of analysis: The current study will adopt interpretative phenomenological analysis to to examine the pain experience of the participants. After data was collected through interview, transcripts will be coded in detail. In the process of analyzing the text, the investigators will categorize the text into themes.

The results of this study can become an important basis for clinical care of patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Individual with non-malignant persistent low back pain that has lasted for at least three months.
* Individual that is willing to undergo interview about their pain experience.
* Individual ages between 20 and 100.

Exclusion Criteria:

* Individual with cognitive or psychological impairments that may compromise the ability to understand the interviewing questionnaire.
* Individual younger that 20 years old.
* The pain is clearly related to spinal cancer.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants should have persistent low back pain that has lasted for at least three months. Pain is a very subjective experience, so it is not necessary that the participant has to be diagnosed by a physician.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain resilience scale (PRS) | 8 weeks
  A 14-item scale used to measure the level of pain resilience. Participant could choose from 0 to 4 on each item to indicate how much one agrees to the statement used to describe one's reaction under persisting pain. "0" indicates "strongly disagree" while "4" indicates "fully agree". Higher total score on the PRS indicates higher resilience to pain.
Spirituality | 8 weeks
  Participant gives a simple yes/no answer as to whether the participant has a religion or participate in religious activities.
Patient Health Questionnaire-9 | 8 weeks
  Patient Health Questionnaire-9 is a 9-item scale used to measure the level of depression in a respondent. Participant chooses from 0 to 3 on each item to indicate the frequency of experiencing each listed symptoms that might be part of depression. Higher total score indicates higher level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Jun Liu, MSc, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Chang-hua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Personal identifiers will be removed before data sharing (if we decide to share the data). Currently, we prefer to share only the descriptive statistics of the demographic data.

REFERENCES:
- [Result] Slepian PM, Ankawi B, Himawan LK, France CR. Development and Initial Validation of the Pain Resilience Scale. J Pain. 2016 Apr;17(4):462-72. doi: 10.1016/j.jpain.2015.12.010. Epub 2015 Dec 31. PMID 26748044
- [Result] Ankawi B, Slepian PM, Himawan LK, France CR. Validation of the Pain Resilience Scale in a Chronic Pain Sample. J Pain. 2017 Aug;18(8):984-993. doi: 10.1016/j.jpain.2017.03.013. Epub 2017 Apr 18. PMID 28428092
- [Result] Gonzalez CE, Okunbor JI, Parker R, Owens MA, White DM, Merlin JS, Goodin BR. Pain-Specific Resilience in People Living With HIV and Chronic Pain: Beneficial Associations With Coping Strategies and Catastrophizing. Front Psychol. 2019 Sep 6;10:2046. doi: 10.3389/fpsyg.2019.02046. eCollection 2019. PMID 31555190
- [Derived] Liu LJ, Peng HL, Lin EM, Liang WP. Do We Ask What the Deities Can Do for Us? The Roles of Dao Religion and Resilience in Suicidality in Chronic Pain. Pain Res Manag. 2025 Apr 17;2025:3056383. doi: 10.1155/prm/3056383. eCollection 2025. PMID 40276019